CLINICAL TRIAL: NCT05715346
Title: A Phase 1/2a Study of LEV102 Topical Gel in Subjects With Acquired Blepharoptosis
Brief Title: LEV102 Topical Gel in Acquired Blepharoptosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Levation Pharma, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LEV102-CS01
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Results first posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Acquired Blepharoptosis
Keywords: Blepharoptosis
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Intervention Model Description: Double-masked parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LEV102 Topical Gel, 2.0% (Experimental)
  Interventions: Drug: LEV102 2.0%
- LEV102 Topical Gel, 1.0% (Experimental)
  Interventions: Drug: LEV102 1.0%
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: LEV102 1.0% — Oxymetazoline ophthalmic gel
  Arms: LEV102 Topical Gel, 1.0%
Drug: LEV102 2.0% — Oxymetazoline ophthalmic gel
  Arms: LEV102 Topical Gel, 2.0%
Drug: Vehicle — Vehicle ophthalmic gel
  Arms: Vehicle

SUMMARY:
Phase 1/2a, multicenter, randomized, vehicle-controlled, double-masked, multiple-dose, parallel-group study conducted in adult subjects with acquired blepharoptosis.

DETAILED DESCRIPTION:
This is a Phase 1/2a, multicenter, randomized, vehicle-controlled, double-masked, single-dose, parallel-group study conducted in adult subjects with acquired blepharoptosis. Subjects will receive a one-time application of randomized, double-masked IP. Approximately 30 subjects will be enrolled in this study. Eligible subjects will be randomized to 1 of the following 3 treatment groups in a 1:1:1 ratio and will receive a single dose of double-masked IP externally on the upper eyelid of both eyes (OU):

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all the following inclusion criteria will be eligible to participate in the study. Subjects must:

1. Be male or female subjects 25 years of age or older at the time of Screening (Visit 1)
2. Have complaints of aesthetically unacceptable upper eyelid position for both eyes making them desirous for elevation, or have complaints of superior visual field defects in both eyes that impact activities of daily living
3. Present with the following at Screening (Visit 1):

   a. At least one eye that meets both of the following criteria: i. Margin Reflex Distance 1 MRD1 ≤2 mm (no visible central pupillary light reflex defaults to 0) ii. Current corrected VA, using subject's own prescription eyeglasses, if applicable, in the qualifying eye(s) of +0.3 LogMAR (Logarithm of the Minimum Angle of Resolution) or better as assessed by ETDRS b. Demonstrate upper eyelid elevation ≥0.5 mm change from baseline in MRD1 in both eyes in response to a single drop of oxymetazoline 0.1% ophthalmic solution)to each eye at Screening
4. Women of Childbearing Potential must agree to use an approved method of birth control from the date they sign the informed consent form (ICF) until after the last study visit (Follow-Up Visit)
5. Be able to give informed consent and willing to comply with all study visits and examinations

Exclusion Criteria:

1. Have any other ocular pathology other than ptosis requiring treatment with topical prescription ophthalmic drops in either eye (e.g., glaucoma, dry eye)
2. Have narrow angles, glaucoma, intraocular pressure >23 mmHg or diagnosis of ocular hypertension, cup-to-disc ratio of >0.7, or history of any glaucoma eye surgery in either eye
3. Have any active ocular or peri-ocular infection; any history of recurrent or chronic infection or inflammation in either eye
4. Have a history of allergic reaction to the investigational drug or any of its components
5. Within 7 days of Screening (Visit 1), or anticipated use during the study, use of any systemic, intranasal, topical dermatologic, or ophthalmic α-adrenergic agonist (including brimonidine) or antagonist including nasal or ocular or oral decongestants including pseudoephedrine, oxymetazoline topical ophthalmic solution, oxymetazoline topical dermatologic cream
6. Subjects who are pregnant or breast-feeding

Ages: 25 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-06-24 (Actual); Study Completion 2023-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Houman D Hemmati, MD PhD, Study Chair — Levation Pharma, Ltd.
Locations (3):
- United States (3):
  - Eye Research Foundation, Newport Beach, California
  - Steve Yoelin Medical Associates, Newport Beach, California
  - Brian Biesman, M.D, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LEV102 Topical Gel, 2.0% | LEV102 Topical Gel, 1.0% | Vehicle
Started | 11 | 11 | 11
Completed | 11 | 11 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEV102 Topical Gel, 2.0% | LEV102 Topical Gel, 1.0% | Vehicle | Total
Number analyzed (Participants) | 11 | 11 | 11 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 4 | 15
  >=65 years | 4 | 7 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (10.3) | 66.3 (15.9) | 65.1 (11.2) | 64.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 8 | 25
  Male | 2 | 3 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 11 | 11 | 10 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Treatment-Emergent Adverse Events [Safety and Tolerability])
Description: Adverse events
Time Frame: Day 2-5
Measure: Count of Participants; unit: Participants
Arm/Group | LEV102 Topical Gel, 2.0% | LEV102 Topical Gel, 1.0% | Vehicle
Number analyzed (Participants) | 11 | 11 | 11
Participants | 0 | 0 | 0

2. Secondary Outcome: Upper Eyelid Height
Description: Percentage of subjects with increase in Margin reflex distance 1 (MRD1) of 1 mm at Hours 2 and 6 on Day 1
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | LEV102 Topical Gel, 2.0% | LEV102 Topical Gel, 1.0% | Vehicle
Number analyzed (Participants) | 11 | 11 | 11
Participants | 7 | 4 | 2

ADVERSE EVENTS:
Time Frame: 2-5 days
Arm/Group | LEV102 Topical Gel, 2.0% | LEV102 Topical Gel, 1.0% | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI to collegially coordinate presentations and papers with Sponsor's scientists.

DOCUMENTS (2):
  • Study Protocol (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT05715346/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT05715346/SAP_001.pdf